CLINICAL TRIAL: NCT07277426
Title: Evaluation of Conjunctival Rotational Flap Compared to Conjunctival Autograft After Surgical Removal of Primary Pterygium: A Randomized Controlled Trial
Brief Title: Comparing Two Surgical Methods to Prevent Pterygium Regrowth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: College of Physicians and Surgeons Pakistan (Other)
Responsible Party: Principal Investigator, Faiz ur rahman, Postgraduate Resident, Department of Operative Dentistry, College of Physicians and Surgeons Pakistan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SGTH-Oph-Pterygium-001
Record Dates: First submitted 2025-11-30; First posted 2025-12-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-11

CONDITIONS: Pterygium
Keywords: Conjunctival Autograft; Conjunctival Rotational Flap; Pterygium Recurrence
MeSH Terms: conditions — Pterygium

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of two parallel groups for the duration of the study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rotational Flap (Experimental): A hinged conjunctival flap created adjacent to the excision site and rotated to cover the scleral defect while maintaining partial vascular attachment.
  Interventions: Procedure: Conjunctival Rotational Flap; Procedure: Conjunctival Autograft
- Conjunctival Autograft (Active Comparator): A free conjunctival graft harvested from the superior bulbar conjunctiva and transplanted to the scleral bed after pterygium excision.
  Interventions: Procedure: Conjunctival Rotational Flap; Procedure: Conjunctival Autograft

INTERVENTIONS:
Procedure: Conjunctival Rotational Flap — A surgical technique where adjacent conjunctival tissue, remaining partially attached, is rotated to cover the exposed sclera after pterygium excision.
Procedure: Conjunctival Autograft — A surgical technique where a free graft of conjunctiva is harvested from the superior bulbar conjunctiva and sutured or glued over the scleral defect after pterygium excision

SUMMARY:
This study compares two surgical techniques for preventing the regrowth of a pterygium, a non-cancerous growth on the eye. After surgically removing the pterygium, surgeons will cover the area with either a flap of nearby tissue that is rotated into place (Rotational Flap) or with a free graft of tissue taken from under the upper eyelid (Autograft). The main goal is to see which method is better at preventing the pterygium from growing back over a 6-month period. A total of 342 patients with a primary pterygium will be randomly assigned to one of the two surgical groups.

DETAILED DESCRIPTION:
This is a single-center, prospective, randomized controlled trial to be conducted at the Department of Ophthalmology, Saidu Group of Teaching Hospital, Swat. The study aims to compare the efficacy of the Conjunctival Rotational Flap versus the Conjunctival Autograft in reducing recurrence rates following primary pterygium excision. Adult patients aged 18-60 with primary pterygium will be enrolled. Participants will be randomly allocated into two groups: Group A (Conjunctival Rotational Flap) and Group B (Conjunctival Autograft). The primary outcome measure is the absence of clinical recurrence, defined as fibrovascular tissue crossing ≥ 1 mm onto the cornea, assessed at the 6-month postoperative follow-up visit via slit-lamp examination. Secondary outcomes may include operative time and postoperative complications. Data will be analyzed using SPSS version 23, with a p-value of ≤ 0.05 considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* • Age 18-60

  * Either gender
  * Primary pterygium

Exclusion Criteria:

* • Collagen vascular disease

  * Autoimmune disorders
  * Pregnancy
  * Ocular surface infection
  * Previous limbal surgery
  * Recurrent or pseudo-pterygium
  * Ocular trauma
  * Corneal opacity/degeneration'

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-07-02 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Pterygium Recurrence Rate | 6 months postoperatively
  Absence of clinical recurrence, defined as a quiet ocular surface with no fibrovascular regrowth ≥ 1 mm onto the cornea, as measured by slit-lamp examination.

IPD SHARING:
Plan to Share IPD: No